CLINICAL TRIAL: NCT04229992
Title: Calcium: Magnesium Balance, Microbiota, and Necroptosis and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Martha Shrubsole, Research Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 100106d; R01DK110166 (NIH); R01CA149633 (NIH)
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — magnesium diglycinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GG genotype and magnesium treatment (Active Comparator): Participants who have the GG genotype will be assigned to magnesium glycinate
  Interventions: Dietary Supplement: Magnesium glycinate
- GG genotype and placebo (Placebo Comparator): Participants who have the GG genotype will be assigned to placebo group
  Interventions: Dietary Supplement: Placebo
- GA/AA genotype and magnesium treatment (Active Comparator): Participants who have the GA/AA genotype will be assigned to magnesium glycinate
  Interventions: Dietary Supplement: Magnesium glycinate
- GA/AA genotype and Placebo (Placebo Comparator): Participants who have the GA/AA genotype will be assigned to placebo group
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium glycinate — Oral administration of magnesium glycinate daily for 12 weeks
  Arms: GA/AA genotype and magnesium treatment; GG genotype and magnesium treatment
Dietary Supplement: Placebo — Oral administration of identical-appearing placebo daily for 12 weeks
  Arms: GA/AA genotype and Placebo; GG genotype and placebo

SUMMARY:
Transient receptor potential melastatin 7 (TRPM7), a magnesium (Mg) -regulated chanzyme possessing both ion channel and kinase activities, has a much stronger affinity to Mg2+ than calcium (Ca)2+. We previously reported that individuals with the TRPM7 GA/AA genotype and consumed diets high in Ca:Mg ratio had an increased risk of colorectal polyps. The TRPM7 gene was also observed to possess "driver" mutations that contribute to developing multiple cancers. However, the molecular mechanism remains unclear.

To identify if the gut microbiota plays a role in this association, we will investigate whether optimizing Ca:Mg intake ratios to 2.3 altered the abundance of the microbes (e.g. associated with TRPM7 genotype and the risk of metachronous polyps) at the genus level in at least one sample type among stool, swab and tissue in a double-blind 2x2 factorial (TRPM7 genotype and Ca:Mg ratios) randomized trial (Personalized Prevention of Colorectal Cancer Trial, NCT01105169).

ELIGIBILITY:
Inclusion Criteria:

• Participants from the parent study (Personalized Prevention of Colorectal Cancer Trial, NCT#01105169, IRB#100106)

Exclusion Criteria:

• Participants did not provide any stool/swab/rectal biopsy sample in the parent study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Shrubsole, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Sun E, Zhu X, Ness RM, Murff HJ, Sun S, Yu C, Fan L, Azcarate-Peril MA, Shrubsole MJ, Dai Q. Magnesium treatment increases gut microbiome synthesizing vitamin D and inhibiting colorectal cancer: results from a double-blind precision-based randomized placebo-controlled trial. Am J Clin Nutr. 2025 Nov;122(5):1185-1194. doi: 10.1016/j.ajcnut.2025.09.011. Epub 2025 Sep 12. PMID 40946805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants, aged 40-85 y, with colorectal polyp or polyp-free individuals with high risk of colorectal cancer and had a calcium intake of ≥700 and <2000 mg/d, and their calcium-to-magnesium intake ratio was >2.6 (based on baseline two 24-hour dietary recalls) and have blood samples were recruited from Vanderbilt patient sources from March 11, 2011 to Jan 30, 2016 .
Groups:
- GG Genotype and Magnesium Treatment: Participants who have the GG genotype were assigned to magnesium glycinate
  Magnesium glycinate: Oral administration of magnesium glycinate daily for 12 weeks
- GG Genotype and Placebo: Participants who have the GG genotype were assigned to placebo group
  Placebo: Oral administration of identical-appearing placebo daily for 12 weeks
- GA/AA Genotype and Magnesium Treatment: Participants who have the GA/AA genotype were assigned to magnesium glycinate
  Magnesium glycinate: Oral administration of magnesium glycinate daily for 12 weeks
- GA/AA Genotype and Placebo: Participants who have the GA/AA genotype were assigned to placebo group
  Placebo: Oral administration of identical-appearing placebo daily for 12 weeks
Period: Overall Study
Arm/Group | GG Genotype and Magnesium Treatment | GG Genotype and Placebo | GA/AA Genotype and Magnesium Treatment | GA/AA Genotype and Placebo
Started | 77 | 78 | 47 | 48
Completed | 76 | 75 | 43 | 45
Not Completed | 1 | 3 | 4 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GG Genotype and Magnesium Treatment | GG Genotype and Placebo | GA/AA Genotype and Magnesium Treatment | GA/AA Genotype and Placebo | Total
Number analyzed (Participants) | 76 | 75 | 43 | 45 | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 52 | 29 | 26 | 160
  >=65 years | 23 | 23 | 14 | 19 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (8.2) | 60.0 (8.5) | 60.0 (7.0) | 61.4 (7.6) | 60.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 35 | 23 | 23 | 113
  Male | 44 | 40 | 20 | 22 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 0 | 3
  White | 74 | 74 | 43 | 45 | 236
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 76 | 75 | 43 | 45 | 239

OUTCOME MEASURES:

1. Primary Outcome: Comparisons of the Changes of Genera Prevotella by Mg Treatment vs. Placebo in Rectal Mucosa, Swab and Stool Samples
Description: changes=value at 12 weeks minus value at baseline. Difference between post-treatment and baseline, means increase or reduced the abundance of genera Prevotella in the test samples (rectal mucosa or rectal swab or stool).
Time Frame: 12 weeks
Population: Among participants with with rectal mucosa and rectal swab and stool samples.
Measure: Mean (Standard Error); unit: percentage of sample
Arm/Group | GG Genotype and Magnesium Treatment | GG Genotype and Placebo | GA/AA Genotype and Magnesium Treatment | GA/AA Genotype and Placebo
Number analyzed (Participants) | 73 | 70 | 42 | 44
percentage of sample
  Rectal Mucosa | 0.108 (2.268) | 0.245 (2.686) | -0.076 (2.355) | 0.132 (2.034)
  Rectal Swab | -0.174 (1.954) | -0.095 (2.239) | -0.919 (2.165) | 0.364 (2.111)
  Stool | -0.059 (1.716) | -0.001 (1.814) | 0.363 (1.276) | 0.137 (1.639)
Statistical Analysis 1: Comparison: GG Genotype and Magnesium Treatment vs GG Genotype and Placebo vs GA/AA Genotype and Magnesium Treatment vs GA/AA Genotype and Placebo; 1. GG genotype and magnesium treatment vs GG genotype and placebo; 2. GA/AA genotype and magnesium treatment vs GA/AA genotype and Placebo; Test type: Superiority; p < 0.05, Regression, Linear; P value was calculated using general linear mode adjusted for age, sex, BMI and baseline level

2. Primary Outcome: Comparisons of the Changes of Genera Bacteroides by Mg Treatment vs. Placebo in Rectal Mucosa, Swab and Stool Samples
Description: as for outcome 1
Time Frame: 12 weeks
Population: Among participants with with rectal mucosa and rectal swab and stool samples.
Measure: Mean (Standard Error); unit: percentage of sample
Arm/Group | GG Genotype and Magnesium Treatment | GG Genotype and Placebo | GA/AA Genotype and Magnesium Treatment | GA/AA Genotype and Placebo
Number analyzed (Participants) | 73 | 70 | 42 | 44
percentage of sample
  Rectal mucosa | -0.030 (0.205) | -0.027 (0.252) | 0.039 (0.208) | -0.025 (0.196)
  Rectal swab | 0.024 (0.413) | -0.013 (0.465) | -0.041 (0.355) | -0.017 (0.283)
  Stool | -0.063 (0.536) | 0.022 (0.410) | -0.105 (0.377) | 0.084 (0.418)
Statistical Analysis 1: Comparison: GG Genotype and Magnesium Treatment vs GG Genotype and Placebo vs GA/AA Genotype and Magnesium Treatment vs GA/AA Genotype and Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, Regression, Linear; P value was calculated using general linear mode adjusted for age, sex, BMI and baseline level

ADVERSE EVENTS:
Time Frame: In the 12 weeks trial, we conducted safety and compliance calls to collect adverse event data.
Description: The definition of adverse event and/or serious adverse event is from the clinicaltrials.gov Definitions.
  We conducted safety and compliance calls to collect adverse event data.
Arm/Group | GG Genotype and Magnesium Treatment | GG Genotype and Placebo | GA/AA Genotype and Magnesium Treatment | GA/AA Genotype and Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/78 | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/78 | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 1/77 | 2/78 | 3/47 | 1/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GG Genotype and Magnesium Treatment (N=77) | GG Genotype and Placebo (N=78) | GA/AA Genotype and Magnesium Treatment (N=47) | GA/AA Genotype and Placebo (N=48)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bleeding after the rectal biopsy procedure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feel sick (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Having an adverse effect on his blood pressure medication (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0
Weight gain, migraine and swelling with arthritic pain in fingers (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT04229992/Prot_SAP_000.pdf